CLINICAL TRIAL: NCT01519037
Title: Evaluation of the Interaction Between a Calcimimetic Agent (Cinacalcet) and the Renin Angiotensine Aldosterone System in Healthy Volunteers
Brief Title: Interaction Between a Calcimimetic Agent and the Renin Angiotensine Aldosterone System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Michel Burnier, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2011DR4219
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Relationship Between Calcimimetic and the RAAS
Keywords: calcimimetic agent; RAAS; renin; aldosterone
MeSH Terms: interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcimimetic agent (cinacalcet) (Active Comparator): 3 days of a low-sodium diet (50 mmol of Na+ per day, equivalent to 3 grams of salt/day), followed by an investigation day at the hospital during which the subjects will be studied before and after exposure to the cinacalcet or the placebo. The 2 periods will be separated by a therapeutic wash-out lasting 14-28 days. The total length of the study per participant will be 1, max. 2 months
  Interventions: Drug: Cinacalcet 60 MG
- Placebo (Placebo Comparator): 3 days of a low-sodium diet (50 mmol of Na+ per day, equivalent to 3 grams of salt/day), followed by an investigation day at the hospital during which the subjects will be studied before and after exposure to the cinacalcet or placebo. The 2 periods will be separated by a therapeutic wash-out lasting 14-28 days. The total length of the study per participant will be 1, max. 2 months
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Cinacalcet 60 MG — one dose of oral cinacalcet, 60mg
  Arms: calcimimetic agent (cinacalcet)
Drug: Placebo oral tablet — one tablet of placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate, in healthy volunteers, the acute modulating effect of cinacalcet on the RAAS, the effect of furosemide on parathyroid secretion of PTH and the interaction between furosemide and cinacalcet on parathyroid hormone secretion.

DETAILED DESCRIPTION:
The clinical trial will be monocentric (Service of Nephrology and Hypertension at CHUV, Lausanne) and will include 24 patients. The volunteers will get involved after inclusion (Inclusion Visit) in a crossover study over two double-blind periods. The order of the two periods (placebo or cinacalcet) will be randomized. Each period comprises 3 days of a low-sodium diet (50 mmol of Na+ per day, equivalent to 3 grams of salt/day), followed by an investigation day at the hospital during which the subjects will be studied before and after exposure to the cinacalcet or placebo. The 2 periods will be separated by a therapeutic wash-out lasting 14-28 days. The total length of the study per participant will be 1, max. 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Male

  * Age > 18 and < 45 years old
  * Caucasian
  * Non-smoker
  * BMI >18 and < 25 Kg/m2
  * Normal clinical examination
  * ECG normal, 12 leads
  * Systolic arterial pressure (SBP) ≥100 ≤ 139 mmHg and diastolic arterial pressure (DBP) ≥50 ≤ 89 mmHg (after 5 minutes lying down, 3 measurements at 2-minute intervals; Omron machine; left arm)
  * Heart rate (HR) ≥ 45 ≤ 90 beats/min
  * Subject capable of understanding the written information and the written consent form.
  * Subject must have given written, dated and signed consent before starting any trial procedure.

Exclusion Criteria:

* • Female

  * Age < 18 or > 45 years old
  * Electrolyte disturbances, defined as any sodium, potassium, total or ionized calcium, phosphate or magnesium value outside of the laboratory's reference values (at the Inclusion Visit).
  * Seropositive for HIV, HBV or HCV (at the Inclusion Visit).
  * Positive detection of drugs in urine (opiates, cannabinoids, cocaine, benzodiazepines, amphetamines or barbiturates) (at the Inclusion Visit).
  * Fall in SBP > or DBP > 10 mmHg after standing for 1 minute or any clinical manifestation of postural hypotension (at the Inclusion Visit).
  * Any history of diseases or clinically significant conditions which may be gastrointestinal (such as gastritis or gastric ulcer), respiratory, psychiatric, neurological (medical history of convulsions), renal, hepatic or cardiac or other diseases/conditions or abnormal physical signs which may interfere with the study's objectives. The investigator may disqualify any subject for a valid medical or psychiatric reason.
  * Ongoing involvement or in the 60 days prior to the Inclusion Visit in another research study.
  * Chronic use of any medication (prescribed or not) during the 4 weeks prior to the Inclusion Visit (only the use of medications such as paracetamol for headaches will be tolerated at the lowest dose possible.
  * Use of any medication known as CYP P450 3A4 inhibitors during the 12 weeks prior to the Inclusion Visit (amiodarone, diltiazem, verapamil, ketoconazole, itraconazole, voriconazole, posaconazole, fluconazole, miconazol, ritonavir, nelfinavir, amprenavir, indinavir, atazanavir, erythromycin, clarithromycin, josamycin, telithromycin)
  * Donation of blood, plasma and/or marrow in the 3 months prior to the Inclusion Visit
  * Medical history of dependence on drugs or alcohol abuse as defined by the DSM IVR, criteria for diagnosing drug and alcohol abuse and dependence on drugs.
  * Medical history of intolerant reactions to cinacalcet or furosemide (or derivatives of sulfamides)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effect of cinacalcet compared to placebo on plasma renin activity | up to 36 days
  to determine the acute effect of a single high dose of cinacalcet compared to placebo on plasma renin activity (PRA), under RAAS-stimulating conditions (low sodium diet, furosemide injection) by PRA plasma measure

SECONDARY OUTCOMES:
effect of cinacalcet administered as single dose (compared to placebo) on plasma aldosterone and on hemodynamics | up to 36 days
  to determine the effect of cinacalcet administered as single dose (compared to placebo) on plasma aldosterone and on hemodynamics (blood pressure, heart rate), under RAAS stimulating conditions (low sodium diet, furosemide injection).

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, Professor, Principal Investigator — CHUV
Locations (1):
- CHUV, service de néphrologie/hypertension, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Background] Maillard MP, Tedjani A, Perregaux C, Burnier M. Calcium-sensing receptors modulate renin release in vivo and in vitro in the rat. J Hypertens. 2009 Oct;27(10):1980-7. doi: 10.1097/HJH.0b013e32832f0d22. PMID 19593209
- [Result] Muller ME, Forni Ogna V, Maillard M, Stoudmann C, Zweiacker C, Anex C, Wuerzner G, Burnier M, Bonny O. Furosemide stimulation of parathormone in humans: role of the calcium-sensing receptor and the renin-angiotensin system. Pflugers Arch. 2015 Dec;467(12):2413-21. doi: 10.1007/s00424-015-1714-4. Epub 2015 Jun 20. PMID 26089029